CLINICAL TRIAL: NCT02312297
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single-dose, Crossover, Bioequivalence Study Comparing Minocycline Hydrochloride 135 mg Extended Release Tablets (Containing Minocycline Hydrochloride 135 mg) of OHM Laboratories, USA (A Subsidiary of Ranbaxy Pharmaceuticals Inc. USA) With SolodynTM Extended Release Tablets (Containing Minocycline Hydrochloride 135 mg) of AAI Pharma, Inc. in Healthy, Adult, Male, Human Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Minocycline HCl 135 mg ER Tablet Sunder Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 237_MINOC_08
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Minocycline hydrochloride extended release tablets 135 mg
  Interventions: Drug: Minocycline hydrochloride
- Reference (Active Comparator): Solodyn Extended Release Tablets 135 mg
  Interventions: Drug: Minocycline hydrochloride

INTERVENTIONS:
Drug: Minocycline hydrochloride — extended release tablets 135 mg

SUMMARY:
The study was conducted as an open-label, balanced, randomized, two-treatment, two-period, two-sequence, single-dose, crossover, bioequivalence study comparing Minocycline hydrochloride extended release tablets 135 mg manufactured by OHM Laboratories Inc. with SolodynTM extended release tablets 135 mg manufactured by AAI Pharma, Inc Wilmington, NC 28405 and manufactured for Medicis, The Dermatology Company Scottsdale, AZ 85258 in healthy, adult, male, human subjects under fasting condition.

DETAILED DESCRIPTION:
Test for drugs of abuse (opiates and cannabinoids) in urine and breath test for alcohol were carried out prior to admission in each period of the study. Following an overnight fast of at least 10 hour, a single oral dose of minocycline hydrochloride extended release tablet 135 mg of either test or reference formulation was administered during each period of the study, along with 240 mL of drinking water at ambient temperature under low light condition and under supervision of trained study personnel.

During the course of the study, safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical parameters, serology and urine analysis) at baseline. Adverse event monitoring was done throughout the study. Laboratory parameters of hematology and biochemistry (except blood glucose and cholesterol) were repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Volunteers who met the following criteria were included in the study

1. Were in the age range of 18-45 years
2. Were neither overweight nor underweight for their height as per the Life Insurance Corporation of India height/weight chart for non-medical cases
3. Had voluntarily given written informed consent to participate in this study
4. Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study
5. Male subjects and:

   * Whose female partner(s) was/were not pregnant or was/were not planning to become pregnant
   * Whose female partner(s) was/were using at least one highly effective and one acceptable method of birth control (at the same time) for the duration of the study and for 2 weeks after completion of the study, such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence. Dual method of contraception must be used during the study and for 2 weeks after its discontinuation
   * Whose female partner was surgically sterile (bilateral tubal ligation, bilateral oophorectomy, hysterectomy)
   * Those using condoms even if vasectomy has been done; during the study and for 2 weeks after completion of the study

Exclusion Criteria:

1. Hypersensitivity to minocycline or related group of drugs or to any other drug
2. History of diarrhoea in last one week or antibiotic induced diarrhoea
3. Frequent episodes of light headedness, vertigo and dizziness preceding one week
4. History of photosensitivity
5. Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations
6. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma, head-injury or coma
7. History of any psychiatric illness, which may impair the ability to provide written informed consent
8. Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection
9. Presence of values which are out of acceptable limits for haemoglobin, total white blood cells count, differential WBC count or platelet count
10. Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
11. Presence of values which are out of acceptable limits for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol
12. Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (> 4/HPF), glucose (positive) or protein (positive)
13. Clinically abnormal ECG or Chest X-ray
14. Regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period
15. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period
16. Use of any enzyme modifying drugs within 30 days prior to Day 1 of this study
17. Participation in any clinical trial within 12 weeks preceding Day 1 of this study
18. Subjects who, through completion of this study, would have donated and /or lost more than 350 ml of blood in the past 3 months other than study participation

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of Minocycline | 0-96 hrs
Peak Plasma Concentration (Cmax) of Minocycline | 0-96 hrs

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm